CLINICAL TRIAL: NCT01953328
Title: A Double-blind, Randomized, Placebo-controlled, Multicenter Study to Evaluate Safety, Tolerability and Efficacy of Evolocumab (AMG 145) on LDL-C in Combination With Statin Therapy in Japanese Subjects With High Cardiovascular Risk and With Hyperlipidemia or Mixed Dyslipidemia
Brief Title: Study of Low-Density Lipoprotein Cholesterol (LDL-C) Reduction Using Evolocumab (AMG 145) in Japanese Patients With Advanced Cardiovascular Risk
Acronym: AMG145
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20120122
Record Dates: First submitted 2013-09-26; First posted 2013-09-30 (Estimated); Results first posted 2015-12-23 (Estimated); Last update posted 2015-12-23 (Estimated); Status verified 2015-11

CONDITIONS: Hyperlipidemia or Mixed Dyslipidemia at High Risk for Cardiovascular Events
Keywords: Japanese, high cholesterol, LDL-C, High Cardiovascular Risk
MeSH Terms: conditions — Hyperlipidemias; Hypercholesterolemia | interventions — Atorvastatin; evolocumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- A5 Placebo Q2W (Placebo Comparator): Participants received atorvastatin 5 mg (A5) once daily during the 4 week lipid stabilization period and then in combination with placebo subcutaneous injection once every 2 weeks (Q2W) for 12 weeks.
  Interventions: Drug: Atorvastatin; Other: Placebo to Evolocumab
- A5 Placebo QM (Placebo Comparator): Participants received atorvastatin 5 mg a day during the 4-week lipid stabilization period and then in combination with placebo subcutaneous injection once every month (QM) for 12 weeks.
  Interventions: Drug: Atorvastatin; Other: Placebo to Evolocumab
- A5 Evolocumab Q2W (Experimental): Participants received atorvastatin 5 mg a day during the 4-week lipid stabilization period and then in combination with 140 mg evolocumab by subcutaneous injection once every 2 weeks for 12 weeks.
  Interventions: Drug: Atorvastatin; Biological: Evolocumab
- A5 Evolocumab QM (Experimental): Participants received atorvastatin 5 mg a day during the 4-week lipid stabilization period and then in combination with 420 mg evolocumab by subcutaneous injection once a month for 12 weeks.
  Interventions: Drug: Atorvastatin; Biological: Evolocumab
- A20 Placebo Q2W (Placebo Comparator): Participants received atorvastatin 20 mg (A20) once daily during the 4 week lipid stabilization period and then in combination with placebo subcutaneous injection once every 2 weeks for 12 weeks.
  Interventions: Drug: Atorvastatin; Other: Placebo to Evolocumab
- A20 Placebo QM (Other): Participants received atorvastatin 20 mg a day during the 4-week lipid stabilization period and then in combination with placebo subcutaneous injection once every month for 12 weeks.
  Interventions: Drug: Atorvastatin; Other: Placebo to Evolocumab
- A20 Evolocumab Q2W (Experimental): Participants received atorvastatin 20 mg a day during the 4-week lipid stabilization period and then in combination with 140 mg evolocumab by subcutaneous injection once every 2 weeks for 12 weeks.
  Interventions: Drug: Atorvastatin; Biological: Evolocumab
- A20 Evolocumab QM (Experimental): Participants received atorvastatin 20 mg a day during the 4-week lipid stabilization period and then in combination with 420 mg evolocumab by subcutaneous injection once a month for 12 weeks.
  Interventions: Drug: Atorvastatin; Biological: Evolocumab

INTERVENTIONS:
Drug: Atorvastatin — Administered orally once a day
  Other Names: Lipitor
Biological: Evolocumab — Administered by subcutaneous injection
  Other Names: AMG 145; Repatha
  Arms: A20 Evolocumab Q2W; A20 Evolocumab QM; A5 Evolocumab Q2W; A5 Evolocumab QM
Other: Placebo to Evolocumab — Administered by subcutaneous injection
  Arms: A20 Placebo Q2W; A20 Placebo QM; A5 Placebo Q2W; A5 Placebo QM

SUMMARY:
The primary objective of the study was to evaluate the effect of 12 weeks of subcutaneous evolocumab administered every 2 weeks and once a month, compared with placebo, on percent change from baseline in LDL-C when used in combination with statin therapy in adults with high cardiovascular risk and with hyperlipidemia or mixed dyslipidemia.

DETAILED DESCRIPTION:
After a screening and placebo run-in period, eligible patients were randomized in a 1:1 ratio to 1 of 2 open-label background statin treatments (atorvastatin 5 mg or 20 mg daily [QD]) and entered a 4-week lipid stabilization period. After the lipid stabilization period, eligible patients were randomized in a 1:1:1:1 ratio to investigational product (evolocumab or placebo) for the 12-week treatment period.

Both randomizations were stratified by subject diagnosis and lipid-lowering therapy as follows:

* current or prior diagnosis of heterozygous familial hypercholesterolemia (HeFH)
* no diagnosis of HeFH and receiving intensive lipid-lowering therapy
* no diagnosis of HeFH and receiving non-intensive lipid-lowering therapy. A participant was considered randomized into the study after successfully completing the screening period, meeting all inclusion/exclusion criteria including meeting final laboratory safety criteria, and undergoing both randomization procedures.

ELIGIBILITY:
Inclusion Criteria: Male or female, Japanese adult, 20-85 years of age; Subjects on stable dose of statin for greater than equal to 4 weeks; Fasting LDL-C greater than equal to 100 mg/dL; Fasting triglycerides less than equal to 400 mg/dL; Subject is at high risk for cardiovascular events. Exclusion Criteria: New York heart Association (NYHA) III or IV - heart failure; Uncontrolled cardiac arrhythmia; Uncontrolled hypertension; Type 1 diabetes, poorly controlled type 2 diabetes; Uncontrolled hypothyroidism or hyperthyroidism

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 409 (Actual)
Dates: Start 2013-10; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (38):
- Japan (38):
  - Research Site, Akita, Akita
  - Research Site, Noda, Chiba
  - Research Site, Fukuoka, Fukuoka
  - Research Site, Kitakyusyu-shi, Fukuoka
  - Research Site, Koriyama-shi, Fukushima
  - Research Site, Maebashi, Gunma
  - Research Site, Takasaki-shi, Gunma
  - Research Site, Sapporo, Hokkaido
  - Research Site, Tsuchiura-shi, Ibaraki
  - Research Site, Hanamaki-shi, Iwate
  - Research Site, Morioka, Iwate
  - Research Site, Takamatsu, Kagawa-ken
  - Research Site, Yokohama, Kanagawa
  - Research Site, Kyoto, Kyoto
  - Research Site, Sendai, Miyagi
  - Research Site, Tomigusuku-shi, Okinawa
  - Research Site, Urasoe-shi, Okinawa
  - Research Site, Ibaraki-shi, Osaka
  - Research Site, Osaka, Osaka
  - Research Site, Toyonaka-shi, Osaka
  - Research Site, Koshigaya-shi, Saitama
  - Research Site, Kumagaya-shi, Saitama
  - Research Site, Niiza-shi, Saitama
  - Research Site, Arakawa-ku, Tokyo
  - Research Site, Chiyoda-ku, Tokyo
  - Research Site, Chofu-shi, Tokyo
  - Research Site, Chuo-ku, Tokyo
  - Research Site, Edogawa-ku, Tokyo
  - Research Site, Hachioji-shi, Tokyo
  - Research Site, Itabashi-ku, Tokyo
  - Research Site, Katsushika-ku, Tokyo
  - Research Site, Koto-ku, Tokyo
  - Research Site, Minato-ku, Tokyo
  - Research Site, Ōta-ku, Tokyo
  - Research Site, Setagaya-ku, Tokyo
  - Research Site, Shibuya-ku, Tokyo
  - Research Site, Shinagawa-ku, Tokyo
  - Research Site, Toshima-ku, Tokyo

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Japanese men and women ≥ 20 to ≤ 85 years of age, with fasting low-density lipoprotein cholesterol (LDL-C) ≥ 100 mg/dL (2.6 mmol/L), fasting triglycerides ≤ 400 mg/dL (4.5 mmol/L), and at high risk for cardiovascular events were eligible to participate. First patient enrolled on 07 October 2013 and last patient enrolled on 17 February 2014.
Pre-assignment Details: 409 participants were randomized to 1 of 2 open-label atorvastatin cohorts (5 mg or 20 mg) for the lipid stabilization period; 404 were then randomized to blinded investigational product. Both randomizations were stratified by heterozygous familial hypercholesterolemia (HeFH) diagnosis and lipid-lowering therapy.
Groups:
- A5 Placebo Q2W: Participants received atorvastatin 5 mg (A5) daily during the 4 week lipid stabilization period and then in combination with placebo subcutaneous injection once every 2 weeks (Q2W) for 12 weeks.
- A5 Placebo QM: Participants received atorvastatin 5 mg daily during the 4-week lipid stabilization period and then in combination with placebo subcutaneous injection once every month (QM) for 12 weeks.
- A5 Evolocumab Q2W: Participants received atorvastatin 5 mg daily during the 4-week lipid stabilization period and then in combination with 140 mg evolocumab by subcutaneous injection once every 2 weeks for 12 weeks.
- A5 Evolocumab QM: Participants received atorvastatin 5 mg daily during the 4-week lipid stabilization period and then in combination with 420 mg evolocumab by subcutaneous injection once a month for 12 weeks.
- A20 Placebo Q2W: Participants received atorvastatin 20 mg (A20) daily during the 4 week lipid stabilization period and then in combination with placebo subcutaneous injection once every 2 weeks for 12 weeks.
- A20 Placebo QM: Participants received atorvastatin 20 mg daily during the 4-week lipid stabilization period and then in combination with placebo subcutaneous injection once every month for 12 weeks.
- A20 Evolocumab Q2W: Participants received atorvastatin 20 mg daily during the 4-week lipid stabilization period and then in combination with 140 mg evolocumab by subcutaneous injection once every 2 weeks for 12 weeks.
- A20 Evolocumab QM: Participants received atorvastatin 20 mg daily during the 4-week lipid stabilization period and then in combination with 420 mg evolocumab by subcutaneous injection once a month for 12 weeks.
Period: Overall Study
Arm/Group | A5 Placebo Q2W | A5 Placebo QM | A5 Evolocumab Q2W | A5 Evolocumab QM | A20 Placebo Q2W | A20 Placebo QM | A20 Evolocumab Q2W | A20 Evolocumab QM
Started | 49 | 50 | 50 | 50 | 52 | 51 | 51 | 51
Received Treatment | 49 | 50 | 50 | 50 | 52 | 51 | 51 | 51
Completed | 49 | 50 | 50 | 50 | 50 | 51 | 51 | 51
Not Completed | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set (all randomized participants who reveid at least 1 dose of blinded investigational product).
Groups:
- Total: Total of all reporting groups
Arm/Group | A5 Placebo Q2W | A5 Placebo QM | A5 Evolocumab Q2W | A5 Evolocumab QM | A20 Placebo Q2W | A20 Placebo QM | A20 Evolocumab Q2W | A20 Evolocumab QM | Total
Number analyzed (Participants) | 49 | 50 | 50 | 50 | 52 | 51 | 51 | 51 | 404
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.1 (9.9) | 60.6 (9.9) | 65.2 (7.8) | 60.1 (11.6) | 60.4 (10.4) | 60.4 (10.5) | 60.1 (9.9) | 61.8 (11.9) | 61.3 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 15 | 23 | 18 | 24 | 18 | 16 | 24 | 160
  Male | 27 | 35 | 27 | 32 | 28 | 33 | 35 | 27 | 244
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 49 | 50 | 50 | 50 | 52 | 51 | 51 | 51 | 404
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stratification Factor [Number; unit: participants] — Intensive statin use was defined as daily atorvastatin ≥ 10 mg, fluvastatin ≥ 80 mg, lovastatin ≥ 40 mg, pitavastatin ≥ 2 mg, pravastatin ≥ 40 mg, rosuvastatin ≥ 5 mg, simvastatin ≥ 20 mg, or any statin plus ezetimibe. Non-intensive is defined as any dose of a statin at least weekly for the last 4 weeks prior to screening and not included in the above.
  participants
    Diagnosis of HeFH | 3 | 2 | 2 | 3 | 3 | 2 | 3 | 3 | 21
    Non-HeFH and Intensive Statin Use | 10 | 10 | 11 | 10 | 11 | 11 | 11 | 11 | 85
    Non-HeFH and Non-Intensive Statin Use | 36 | 38 | 37 | 37 | 38 | 38 | 37 | 37 | 298
LDL-C Concentration [Mean (Standard Deviation); unit: mg/dL] — Baseline lipid parameters were measured after the lipid-stabilization period and prior to administration of first dose of investigational study drug.
  mg/dL | 115.7 (26.0) | 114.0 (29.2) | 121.9 (44.6) | 118.8 (36.6) | 90.9 (25.5) | 90.7 (20.8) | 95.8 (23.6) | 98.0 (25.6) | 105.5 (32.0)
Non-High-Density Lipoprotein Cholesterol (non-HDL-C) Concentration [Mean (Standard Deviation); unit: mg/dL] | 142.0 (30.4) | 141.2 (31.8) | 151.8 (48.8) | 147.8 (39.6) | 118.2 (28.6) | 117.5 (25.1) | 121.8 (29.8) | 122.7 (29.5) | 132.7 (35.9)
Apolipoprotein B Concentration [Mean (Standard Deviation); unit: mg/dL] | 99.0 (20.0) | 100.6 (20.0) | 105.1 (31.2) | 102.2 (24.7) | 85.7 (18.4) | 82.7 (14.6) | 87.2 (19.1) | 87.7 (19.6) | 93.7 (22.8)
Total Cholesterol Concentration [Mean (Standard Deviation); unit: mg/dL] | 199.5 (30.7) | 199.4 (33.2) | 210.4 (47.9) | 202.5 (38.4) | 177.8 (33.0) | 173.6 (29.2) | 177.7 (26.2) | 179.0 (29.4) | 189.8 (36.3)
Total Cholesterol/HDL-C Ratio [Mean (Standard Deviation); unit: ratio] | 3.618 (0.891) | 3.579 (0.827) | 3.743 (1.186) | 3.933 (1.295) | 3.116 (0.760) | 3.170 (0.612) | 3.392 (1.112) | 3.400 (1.071) | 3.491 (1.018)
Apolipoprotein B/Apolipoprotein A-1 Ratio [Mean (Standard Deviation); unit: ratio] | 0.633 (0.160) | 0.628 (0.152) | 0.643 (0.223) | 0.658 (0.235) | 0.529 (0.118) | 0.524 (0.108) | 0.575 (0.177) | 0.576 (0.176) | 0.595 (0.179)
Lipoprotein(a) Concentration [Median (Inter-Quartile Range); unit: nmol/L] | 35.0 [16.5 to 52.5] | 29.5 [9.0 to 47.0] | 36.0 [16.0 to 69.0] | 36.5 [16.0 to 74.0] | 30.0 [11.0 to 45.0] | 35.0 [11.0 to 57.0] | 33.0 [14.0 to 49.0] | 28.0 [11.0 to 60.0] | 33.0 [13.0 to 57.0]
Triglyceride Concentration [Median (Inter-Quartile Range); unit: mg/dL] | 125.0 [90.0 to 174.0] | 128.5 [99.0 to 164.0] | 125.0 [97.0 to 172.0] | 132.0 [103.0 to 171.0] | 120.0 [91.5 to 187.0] | 120.0 [87.0 to 154.0] | 109.0 [82.0 to 149.0] | 113.0 [95.0 to 137.0] | 121.5 [92.0 to 161.5]
HDL-C Concentration [Mean (Standard Deviation); unit: mg/dL] | 57.5 (13.6) | 58.3 (14.6) | 58.6 (12.7) | 54.7 (13.9) | 59.6 (15.4) | 56.0 (11.3) | 55.9 (14.4) | 56.3 (15.7) | 57.1 (14.0)
Very-Low-Density Lipoprotein Cholesterol (VLDL-C) Concentration [Mean (Standard Deviation); unit: mg/dL] | 26.3 (11.0) | 26.8 (10.2) | 29.2 (14.7) | 29.0 (12.8) | 27.4 (12.0) | 25.1 (9.4) | 24.3 (10.7) | 24.7 (10.3) | 26.6 (11.5)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Low-Density Lipoprotein Cholesterol (LDL-C) at the Mean of Weeks 10 and 12
Time Frame: Baseline and Weeks 10 and 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | A5 Placebo Q2W | A5 Placebo QM | A5 Evolocumab Q2W | A5 Evolocumab QM | A20 Placebo Q2W | A20 Placebo QM | A20 Evolocumab Q2W | A20 Evolocumab QM
Number analyzed (Participants) | 49 | 50 | 50 | 50 | 52 | 51 | 51 | 51
percent change | 0.27 (2.21) | 3.91 (2.09) | -73.70 (2.26) | -69.98 (2.02) | -0.42 (3.26) | -2.67 (2.31) | -74.82 (3.26) | -76.93 (2.24)
Statistical Analysis 1: Comparison: A5 Placebo Q2W vs A5 Evolocumab Q2W; The null hypothesis was that there was no difference in the percent change from baseline at the mean of Weeks 10 and 12 in LDL-C between evolocumab and placebo, and the alternative hypothesis was that a mean difference did exist; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; The model includes treatment group, stratification factor, scheduled visit, and the interaction of treatment group with scheduled visit; LS Mean Treatment Difference = -73.97, 95% CI 2-sided [-78.54 to -69.41], Standard Error of Mean 2.30 — Placebo is the reference
Statistical Analysis 2: Comparison: A5 Placebo QM vs A5 Evolocumab QM; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -72.89, 95% CI 2-sided [-77.22 to -68.57], Standard Error of Mean 2.18 — Placebo is the reference
Statistical Analysis 3: Comparison: A20 Placebo Q2W vs A20 Evolocumab Q2W; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -74.41, 95% CI 2-sided [-81.21 to -67.61], Standard Error of Mean 3.43 — Placebo is the reference
Statistical Analysis 4: Comparison: A20 Placebo QM vs A20 Evolocumab QM; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -74.27, 95% CI 2-sided [-78.93 to -69.60], Standard Error of Mean 2.35 — Placebo is the reference

2. Primary Outcome: Percent Change From Baseline in Low-Density Lipoprotein Cholesterol (LDL-C) at Week 12
Time Frame: Baseline and Week 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | A5 Placebo Q2W | A5 Placebo QM | A5 Evolocumab Q2W | A5 Evolocumab QM | A20 Placebo Q2W | A20 Placebo QM | A20 Evolocumab Q2W | A20 Evolocumab QM
Number analyzed (Participants) | 49 | 50 | 50 | 50 | 52 | 51 | 51 | 51
percent change | 1.28 (2.43) | 5.29 (2.19) | -73.57 (2.48) | -64.62 (2.12) | 1.39 (3.51) | -3.49 (2.67) | -74.46 (3.50) | -70.36 (2.61)
Statistical Analysis 1: Comparison: A5 Placebo Q2W vs A5 Evolocumab Q2W; The null hypothesis was that there was no difference in the percent change from baseline at Week 12 in LDL-C between evolocumab and placebo, and the alternative hypothesis was that a mean difference did exist; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -74.85, 95% CI 2-sided [-80.22 to -69.47], Standard Error of Mean 2.71 — Placebo is the reference
Statistical Analysis 2: Comparison: A5 Placebo QM vs A5 Evolocumab QM; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -69.91, 95% CI 2-sided [-74.60 to -65.23], Standard Error of Mean 2.36 — Placebo is the reference
Statistical Analysis 3: Comparison: A20 Placebo Q2W vs A20 Evolocumab Q2W; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -78.85, 95% CI 2-sided [-83.55 to -68.15], Standard Error of Mean 3.88 — Placebo is the reference
Statistical Analysis 4: Comparison: A20 Placebo QM vs A20 Evolocumab QM; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -66.87, 95% CI 2-sided [-72.88 to -60.87], Standard Error of Mean 3.03 — Placebo is the reference

3. Secondary Outcome: Change From Baseline in LDL-C at the Mean of Weeks 10 and 12
Time Frame: Baseline and Weeks 10 and 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | A5 Placebo Q2W | A5 Placebo QM | A5 Evolocumab Q2W | A5 Evolocumab QM | A20 Placebo Q2W | A20 Placebo QM | A20 Evolocumab Q2W | A20 Evolocumab QM
Number analyzed (Participants) | 49 | 50 | 50 | 50 | 52 | 51 | 51 | 51
mg/dL | -14.8 (4.3) | -2.6 (4.3) | -104.1 (4.4) | -88.9 (4.1) | -8.9 (3.2) | -5.7 (3.7) | -77.6 (3.2) | -77.7 (3.6)
Statistical Analysis 1: Comparison: A5 Placebo Q2W vs A5 Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -89.3, 95% CI 2-sided [-98.4 to -80.2], Standard Error of Mean 4.6 — Placebo is the reference
Statistical Analysis 2: Comparison: A5 Placebo QM vs A5 Evolocumab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -86.3, 95% CI 2-sided [-95.1 to -77.5], Standard Error of Mean 4.4 — Placebo is the reference
Statistical Analysis 3: Comparison: A20 Placebo Q2W vs A20 Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -68.7, 95% CI 2-sided [-75.3 to -62.1], Standard Error of Mean 3.3 — Placebo is the reference
Statistical Analysis 4: Comparison: A20 Placebo QM vs A20 Evolocumab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -72.0, 95% CI 2-sided [-79.5 to -64.6], Standard Error of Mean 3.7 — Placebo is the reference

4. Secondary Outcome: Change From Baseline in LDL-C at Week 12
Time Frame: Baseline and Week 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | A5 Placebo Q2W | A5 Placebo QM | A5 Evolocumab Q2W | A5 Evolocumab QM | A20 Placebo Q2W | A20 Placebo QM | A20 Evolocumab Q2W | A20 Evolocumab QM
Number analyzed (Participants) | 49 | 50 | 50 | 50 | 52 | 51 | 51 | 51
mg/dL | -13.7 (4.6) | -0.4 (4.3) | -104.5 (4.6) | -84.0 (4.2) | -7.7 (3.3) | -6.2 (4.0) | -77.2 (3.3) | -71.7 (3.9)
Statistical Analysis 1: Comparison: A5 Placebo Q2W vs A5 Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -90.8, 95% CI 2-sided [-100.9 to -80.7], Standard Error of Mean 5.1 — Placebo is the reference
Statistical Analysis 2: Comparison: A5 Placebo QM vs A5 Evolocumab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -83.6, 95% CI 2-sided [-92.5 to -74.8], Standard Error of Mean 4.5 — Placebo is the reference
Statistical Analysis 3: Comparison: A20 Placebo Q2W vs A20 Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -69.6, 95% CI 2-sided [-76.5 to -62.6], Standard Error of Mean 3.5 — Placebo is the reference
Statistical Analysis 4: Comparison: A20 Placebo QM vs A20 Evolocumab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -65.5, 95% CI 2-sided [-73.8 to -57.1], Standard Error of Mean 4.2 — Placebo is the reference

5. Secondary Outcome: Percent Change From Baseline in Non-HDL-C at the Mean of Weeks 10 and 12
Time Frame: Baseline and Weeks 10 and 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | A5 Placebo Q2W | A5 Placebo QM | A5 Evolocumab Q2W | A5 Evolocumab QM | A20 Placebo Q2W | A20 Placebo QM | A20 Evolocumab Q2W | A20 Evolocumab QM
Number analyzed (Participants) | 49 | 50 | 50 | 50 | 52 | 51 | 51 | 51
percent change | 0.18 (2.13) | 4.26 (1.86) | -68.48 (2.18) | -61.69 (1.80) | -1.57 (2.45) | -1.79 (1.94) | -69.72 (2.45) | -69.07 (1.88)
Statistical Analysis 1: Comparison: A5 Placebo Q2W vs A5 Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -68.67, 95% CI 2-sided [-73.06 to -64.27], Standard Error of Mean 2.21 — Placebo is the reference
Statistical Analysis 2: Comparison: A5 Placebo QM vs A5 Evolocumab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -65.95, 95% CI 2-sided [-69.74 to -62.16], Standard Error of Mean 1.91 — Placebo is the reference
Statistical Analysis 3: Comparison: A20 Placebo Q2W vs A20 Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -68.14, 95% CI 2-sided [-73.30 to -62.99], Standard Error of Mean 2.60 — Placebo is the reference
Statistical Analysis 4: Comparison: A20 Placebo QM vs A20 Evolocumab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -67.28, 95% CI 2-sided [-71.14 to -63.42], Standard Error of Mean 1.94 — Placebo is the reference

6. Secondary Outcome: Percent Change From Baseline in Non-HDL-C at Week 12
Time Frame: Baseline and Week 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | A5 Placebo Q2W | A5 Placebo QM | A5 Evolocumab Q2W | A5 Evolocumab QM | A20 Placebo Q2W | A20 Placebo QM | A20 Evolocumab Q2W | A20 Evolocumab QM
Number analyzed (Participants) | 49 | 50 | 50 | 50 | 52 | 51 | 51 | 51
percent change | 1.12 (2.30) | 5.55 (2.02) | -67.81 (2.35) | -58.03 (1.96) | -0.07 (2.68) | -2.38 (2.22) | -68.89 (2.67) | -63.27 (2.16)
Statistical Analysis 1: Comparison: A5 Placebo Q2W vs A5 Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -68.93, 95% CI 2-sided [-73.96 to -63.89], Standard Error of Mean 2.54 — Placebo is the reference
Statistical Analysis 2: Comparison: A5 Placebo QM vs A5 Evolocumab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -63.58, 95% CI 2-sided [-67.96 to -59.21], Standard Error of Mean 2.20 — Placebo is the reference
Statistical Analysis 3: Comparison: A20 Placebo Q2W vs A20 Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -68.82, 95% CI 2-sided [-74.79 to -62.86], Standard Error of Mean 3.01 — Placebo is the reference
Statistical Analysis 4: Comparison: A20 Placebo QM vs A20 Evolocumab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -60.89, 95% CI 2-sided [-65.78 to -55.99], Standard Error of Mean 2.47 — Placebo is the reference

7. Secondary Outcome: Percent Change From Baseline in Apolipoprotein B at the Mean of Weeks 10 and 12
Time Frame: Baseline and Weeks 10 and 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | A5 Placebo Q2W | A5 Placebo QM | A5 Evolocumab Q2W | A5 Evolocumab QM | A20 Placebo Q2W | A20 Placebo QM | A20 Evolocumab Q2W | A20 Evolocumab QM
Number analyzed (Participants) | 49 | 50 | 50 | 50 | 52 | 51 | 51 | 51
percent change | -0.32 (1.98) | 0.76 (2.06) | -64.76 (2.03) | -58.47 (1.99) | -4.32 (2.27) | -0.85 (1.90) | -64.38 (2.27) | -64.24 (1.84)
Statistical Analysis 1: Comparison: A5 Placebo Q2W vs A5 Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -64.44, 95% CI 2-sided [-68.49 to -60.39], Standard Error of Mean 2.04 — Placebo is the reference
Statistical Analysis 2: Comparison: A5 Placebo QM vs A5 Evolocumab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -59.24, 95% CI 2-sided [-63.30 to -55.17], Standard Error of Mean 2.05 — Placebo is the reference
Statistical Analysis 3: Comparison: A20 Placebo Q2W vs A20 Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -60.06, 95% CI 2-sided [-64.87 to -55.25], Standard Error of Mean 2.42 — Placebo is the reference
Statistical Analysis 4: Comparison: A20 Placebo QM vs A20 Evolocumab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -63.39, 95% CI 2-sided [-67.15 to -59.62], Standard Error of Mean 1.90 — Placebo is the reference

8. Secondary Outcome: Percent Change From Baseline in Apolipoprotein B at Week 12
Time Frame: Baseline and Week 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | A5 Placebo Q2W | A5 Placebo QM | A5 Evolocumab Q2W | A5 Evolocumab QM | A20 Placebo Q2W | A20 Placebo QM | A20 Evolocumab Q2W | A20 Evolocumab QM
Number analyzed (Participants) | 49 | 50 | 50 | 50 | 52 | 51 | 51 | 51
percent change | 0.74 (2.17) | 2.42 (2.26) | -64.83 (2.22) | -54.80 (2.19) | -2.47 (2.48) | -1.89 (2.17) | -62.83 (2.47) | -58.04 (2.11)
Statistical Analysis 1: Comparison: A5 Placebo Q2W vs A5 Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -65.56, 95% CI 2-sided [-70.34 to -60.79], Standard Error of Mean 2.40 — Placebo is the reference
Statistical Analysis 2: Comparison: A5 Placebo QM vs A5 Evolocumab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -57.23, 95% CI 2-sided [-62.05 to -52.40], Standard Error of Mean 2.43 — Placebo is the reference
Statistical Analysis 3: Comparison: A20 Placebo Q2W vs A20 Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -60.37, 95% CI 2-sided [-65.91 to -54.83], Standard Error of Mean 2.79 — Placebo is the reference
Statistical Analysis 4: Comparison: A20 Placebo QM vs A20 Evolocumab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -56.15, 95% CI 2-sided [-60.92 to -51.39], Standard Error of Mean 2.40 — Placebo is the reference

9. Secondary Outcome: Percent Change From Baseline in Total Cholesterol at the Mean of Weeks 10 and 12
Time Frame: Baseline and Weeks 10 and 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | A5 Placebo Q2W | A5 Placebo QM | A5 Evolocumab Q2W | A5 Evolocumab QM | A20 Placebo Q2W | A20 Placebo QM | A20 Evolocumab Q2W | A20 Evolocumab QM
Number analyzed (Participants) | 49 | 50 | 50 | 50 | 52 | 51 | 51 | 51
percent change | -2.49 (1.81) | 1.09 (1.63) | -48.03 (1.85) | -42.34 (1.58) | -4.21 (1.86) | -2.35 (1.68) | -45.19 (1.86) | -45.49 (1.63)
Statistical Analysis 1: Comparison: A5 Placebo Q2W vs A5 Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -45.54, 95% CI 2-sided [-49.35 to -41.73], Standard Error of Mean 1.92 — Placebo is the reference
Statistical Analysis 2: Comparison: A5 Placebo QM vs A5 Evolocumab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -43.43, 95% CI 2-sided [-46.78 to -40.08], Standard Error of Mean 1.69 — Placebo is the reference
Statistical Analysis 3: Comparison: A20 Placebo Q2W vs A20 Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -40.98, 95% CI 2-sided [-44.88 to -37.08], Standard Error of Mean 1.96 — Placebo is the reference
Statistical Analysis 4: Comparison: A20 Placebo QM vs A20 Evolocumab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -43.14, 95% CI 2-sided [-46.48 to -39.80], Standard Error of Mean 1.68 — Placebo is the reference

10. Secondary Outcome: Percent Change From Baseline in Total Cholesterol at Week 12
Time Frame: Baseline and Week 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | A5 Placebo Q2W | A5 Placebo QM | A5 Evolocumab Q2W | A5 Evolocumab QM | A20 Placebo Q2W | A20 Placebo QM | A20 Evolocumab Q2W | A20 Evolocumab QM
Number analyzed (Participants) | 49 | 50 | 50 | 50 | 52 | 51 | 51 | 51
percent change | -1.70 (1.97) | 2.29 (1.67) | -47.14 (2.01) | -39.06 (1.62) | -3.08 (2.00) | -2.44 (1.81) | -44.04 (1.99) | -40.88 (1.76)
Statistical Analysis 1: Comparison: A5 Placebo Q2W vs A5 Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -45.44, 95% CI 2-sided [-49.83 to -41.05], Standard Error of Mean 2.21 — Placebo is the reference
Statistical Analysis 2: Comparison: A5 Placebo QM vs A5 Evolocumab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -41.34, 95% CI 2-sided [-44.84 to -37.85], Standard Error of Mean 1.76 — Placebo is the reference
Statistical Analysis 3: Comparison: A20 Placebo Q2W vs A20 Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -40.96, 95% CI 2-sided [-45.35 to -36.57], Standard Error of Mean 2.21 — Placebo is the reference
Statistical Analysis 4: Comparison: A20 Placebo QM vs A20 Evolocumab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -38.44, 95% CI 2-sided [-42.26 to -34.62], Standard Error of Mean 1.93 — Placebo is the reference

11. Secondary Outcome: Percent Change From Baseline in the Total Cholesterol/HDL-C Ratio at the Mean of Weeks 10 and 12
Time Frame: Baseline and Weeks 10 and 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | A5 Placebo Q2W | A5 Placebo QM | A5 Evolocumab Q2W | A5 Evolocumab QM | A20 Placebo Q2W | A20 Placebo QM | A20 Evolocumab Q2W | A20 Evolocumab QM
Number analyzed (Participants) | 49 | 50 | 50 | 50 | 52 | 51 | 51 | 51
percent change | 3.77 (2.11) | 3.94 (2.16) | -51.00 (2.16) | -48.71 (2.09) | 1.04 (1.82) | 1.58 (2.04) | -49.79 (1.81) | -48.11 (1.98)
Statistical Analysis 1: Comparison: A5 Placebo Q2W vs A5 Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -54.77, 95% CI 2-sided [-59.37 to -50.17], Standard Error of Mean 2.32 — Placebo is the reference
Statistical Analysis 2: Comparison: A5 Placebo QM vs A5 Evolocumab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -52.66, 95% CI 2-sided [-56.95 to -48.36], Standard Error of Mean 2.17 — Placebo is the reference
Statistical Analysis 3: Comparison: A20 Placebo Q2W vs A20 Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -50.83, 95% CI 2-sided [-54.72 to -46.93], Standard Error of Mean 1.96 — Placebo is the reference
Statistical Analysis 4: Comparison: A20 Placebo QM vs A20 Evolocumab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -49.69, 95% CI 2-sided [-53.74 to -45.64], Standard Error of Mean 2.04 — Placebo is the reference

12. Secondary Outcome: Percent Change From Baseline in the Total Cholesterol/HDL-C Ratio at Week 12
Time Frame: Baseline and Week 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | A5 Placebo Q2W | A5 Placebo QM | A5 Evolocumab Q2W | A5 Evolocumab QM | A20 Placebo Q2W | A20 Placebo QM | A20 Evolocumab Q2W | A20 Evolocumab QM
Number analyzed (Participants) | 49 | 50 | 50 | 50 | 52 | 51 | 51 | 51
percent change | 4.73 (2.36) | 4.33 (2.33) | -50.72 (2.40) | -46.62 (2.26) | 1.84 (2.01) | 0.83 (2.20) | -49.52 (2.00) | -44.61 (2.13)
Statistical Analysis 1: Comparison: A5 Placebo Q2W vs A5 Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -55.45, 95% CI 2-sided [-60.93 to -49.98], Standard Error of Mean 2.76 — Placebo is the reference
Statistical Analysis 2: Comparison: A5 Placebo QM vs A5 Evolocumab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -50.95, 95% CI 2-sided [-55.91 to -46.00], Standard Error of Mean 2.50 — Placebo is the reference
Statistical Analysis 3: Comparison: A20 Placebo Q2W vs A20 Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -51.36, 95% CI 2-sided [-55.93 to -46.80], Standard Error of Mean 2.30 — Placebo is the reference
Statistical Analysis 4: Comparison: A20 Placebo QM vs A20 Evolocumab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -45.44, 95% CI 2-sided [-50.08 to -40.81], Standard Error of Mean 2.33 — Placebo is the reference

13. Secondary Outcome: Percent Change From Baseline in Apolipoprotein B/Apolipoprotein A-1 Ratio at the Mean of Weeks 10 and 12
Time Frame: Baseline and Weeks 10 and 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | A5 Placebo Q2W | A5 Placebo QM | A5 Evolocumab Q2W | A5 Evolocumab QM | A20 Placebo Q2W | A20 Placebo QM | A20 Evolocumab Q2W | A20 Evolocumab QM
Number analyzed (Participants) | 49 | 50 | 50 | 50 | 52 | 51 | 51 | 51
percent change | 0.06 (2.02) | 2.79 (2.37) | -66.41 (2.07) | -61.55 (2.29) | -1.92 (2.30) | 1.54 (2.09) | -65.97 (2.30) | -65.72 (2.02)
Statistical Analysis 1: Comparison: A5 Placebo Q2W vs A5 Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -66.47, 95% CI 2-sided [-70.58 to -62.36], Standard Error of Mean 2.07 — Placebo is the reference
Statistical Analysis 2: Comparison: A5 Placebo QM vs A5 Evolocumab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -64.33, 95% CI 2-sided [-69.01 to -59.66], Standard Error of Mean 2.35 — Placebo is the reference
Statistical Analysis 3: Comparison: A20 Placebo Q2W vs A20 Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -64.05, 95% CI 2-sided [-68.90 to -59.20], Standard Error of Mean 2.44 — Placebo is the reference
Statistical Analysis 4: Comparison: A20 Placebo QM vs A20 Evolocumab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -67.26, 95% CI 2-sided [-71.36 to -63.15], Standard Error of Mean 2.07 — Placebo is the reference

14. Secondary Outcome: Percent Change From Baseline in the Apolipoprotein B/Apolipoprotein A-1 Ratio at Week 12
Time Frame: Baseline and Week 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | A5 Placebo Q2W | A5 Placebo QM | A5 Evolocumab Q2W | A5 Evolocumab QM | A20 Placebo Q2W | A20 Placebo QM | A20 Evolocumab Q2W | A20 Evolocumab QM
Number analyzed (Participants) | 49 | 50 | 50 | 50 | 52 | 51 | 51 | 51
percent change | 0.71 (2.11) | 4.08 (2.62) | -67.59 (2.16) | -58.45 (2.53) | -1.15 (2.47) | 0.06 (2.30) | -65.11 (2.46) | -60.56 (2.23)
Statistical Analysis 1: Comparison: A5 Placebo Q2W vs A5 Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -68.29, 95% CI 2-sided [-72.75 to -63.84], Standard Error of Mean 2.24 — Placebo is the reference
Statistical Analysis 2: Comparison: A5 Placebo QM vs A5 Evolocumab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -62.53, 95% CI 2-sided [-68.11 to -56.94], Standard Error of Mean 2.81 — Placebo is the reference
Statistical Analysis 3: Comparison: A20 Placebo Q2W vs A20 Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -63.97, 95% CI 2-sided [-69.44 to -58.50], Standard Error of Mean 2.75 — Placebo is the reference
Statistical Analysis 4: Comparison: A20 Placebo QM vs A20 Evolocumab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -60.62, 95% CI 2-sided [-65.51 to -55.72], Standard Error of Mean 2.47 — Placebo is the reference

15. Secondary Outcome: Percentage of Participants Who Achieved a Mean LDL-C at Weeks 10 and 12 of Less Than 70 mg/dL
Time Frame: Weeks 10 and 12
Population: Full analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | A5 Placebo Q2W | A5 Placebo QM | A5 Evolocumab Q2W | A5 Evolocumab QM | A20 Placebo Q2W | A20 Placebo QM | A20 Evolocumab Q2W | A20 Evolocumab QM
Number analyzed (Participants) | 49 | 50 | 50 | 50 | 52 | 51 | 51 | 51
percentage of participants | 0.0 (2.02) [0.0 to 7.3] | 0.0 (2.37) [0.0 to 7.3] | 98.0 (2.07) [89.5 to 99.6] | 96.0 (2.29) [86.5 to 98.9] | 22.4 (2.30) [13.0 to 35.9] | 15.7 (2.09) [8.2 to 28.0] | 96.0 (2.30) [86.5 to 98.9] | 98.0 (2.02) [89.7 to 99.7]
Statistical Analysis 1: Comparison: A5 Placebo Q2W vs A5 Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; Based on Cochran-Mantel Haenszel test stratified by the stratification factor (HeFH diagnosis and lipid-lowering therapy); Treatment Difference = 98.0, 95% CI 2-sided [86.8 to 99.6]
Statistical Analysis 2: Comparison: A5 Placebo QM vs A5 Evolocumab QM; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 15, analysis 1]; Treatment Difference = 96.0, 95% CI 2-sided [84.1 to 98.9]
Statistical Analysis 3: Comparison: A20 Placebo Q2W vs A20 Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 15, analysis 1]; Treatment Difference = 73.6, 95% CI 2-sided [57.1 to 83.4]
Statistical Analysis 4: Comparison: A20 Placebo QM vs A20 Evolocumab QM; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 15, analysis 1]; Treatment Difference = 82.4, 95% CI 2-sided [67.5 to 90.0]

16. Secondary Outcome: Percentage of Participants Who Achieved LDL-C < 70 mg/dL at Week 12
Time Frame: Week 12
Population: Full analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | A5 Placebo Q2W | A5 Placebo QM | A5 Evolocumab Q2W | A5 Evolocumab QM | A20 Placebo Q2W | A20 Placebo QM | A20 Evolocumab Q2W | A20 Evolocumab QM
Number analyzed (Participants) | 49 | 50 | 50 | 50 | 52 | 51 | 51 | 51
percentage of participants | 0.0 (2.02) [0.0 to 7.3] | 4.2 (2.37) [1.2 to 14.0] | 98.0 (2.07) [89.3 to 99.6] | 96.0 (2.29) [86.5 to 98.9] | 20.4 (2.30) [11.5 to 33.6] | 20.0 (2.09) [11.2 to 33.0] | 96.0 (2.30) [86.5 to 98.9] | 98.0 (2.02) [89.7 to 99.7]
Statistical Analysis 1: Comparison: A5 Placebo Q2W vs A5 Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 15, analysis 1]; Treatment Difference = 98.0, 95% CI 2-sided [86.7 to 99.6]
Statistical Analysis 2: Comparison: A5 Placebo QM vs A5 Evolocumab QM; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 15, analysis 1]; Treatment Difference = 91.8, 95% CI 2-sided [78.2 to 96.0]
Statistical Analysis 3: Comparison: A20 Placebo Q2W vs A20 Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 15, analysis 1]; Treatment Difference = 75.6, 95% CI 2-sided [59.3 to 85.0]
Statistical Analysis 4: Comparison: A20 Placebo QM vs A20 Evolocumab QM; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 15, analysis 1]; Treatment Difference = 78.0, 95% CI 2-sided [62.6 to 86.9]

17. Secondary Outcome: Percent Change From Baseline in Lipoprotein(a) at the Mean of Weeks 10 and 12
Time Frame: Baseline and Weeks 10 and 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | A5 Placebo Q2W | A5 Placebo QM | A5 Evolocumab Q2W | A5 Evolocumab QM | A20 Placebo Q2W | A20 Placebo QM | A20 Evolocumab Q2W | A20 Evolocumab QM
Number analyzed (Participants) | 49 | 50 | 50 | 50 | 52 | 51 | 51 | 51
percent change | 5.23 (6.18) | 4.07 (4.95) | -45.97 (6.27) | -45.01 (4.78) | 6.52 (4.81) | -5.62 (5.00) | -43.03 (4.81) | -49.55 (4.85)
Statistical Analysis 1: Comparison: A5 Placebo Q2W vs A5 Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -51.20, 95% CI 2-sided [-63.88 to -38.52], Standard Error of Mean 6.39 — Placebo is the reference
Statistical Analysis 2: Comparison: A5 Placebo QM vs A5 Evolocumab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -49.08, 95% CI 2-sided [-58.89 to -39.27], Standard Error of Mean 4.94 — Placebo is the reference
Statistical Analysis 3: Comparison: A20 Placebo Q2W vs A20 Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -49.55, 95% CI 2-sided [-59.74 to -39.35], Standard Error of Mean 5.14 — Placebo is the reference
Statistical Analysis 4: Comparison: A20 Placebo QM vs A20 Evolocumab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -43.93, 95% CI 2-sided [-53.75 to -34.12], Standard Error of Mean 4.95 — Placebo is the reference

18. Secondary Outcome: Percent Change From Baseline in Lipoprotein(a) at Week 12
Time Frame: Baseline and Week 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | A5 Placebo Q2W | A5 Placebo QM | A5 Evolocumab Q2W | A5 Evolocumab QM | A20 Placebo Q2W | A20 Placebo QM | A20 Evolocumab Q2W | A20 Evolocumab QM
Number analyzed (Participants) | 49 | 50 | 50 | 50 | 52 | 51 | 51 | 51
percent change | 4.35 (6.86) | 7.03 (5.47) | -45.72 (6.93) | -41.74 (5.29) | 10.75 (5.15) | -5.73 (5.18) | -41.93 (5.13) | -45.70 (5.02)
Statistical Analysis 1: Comparison: A5 Placebo Q2W vs A5 Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -50.07, 95% CI 2-sided [-65.25 to -34.90], Standard Error of Mean 7.64 — Placebo is the reference
Statistical Analysis 2: Comparison: A5 Placebo QM vs A5 Evolocumab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -48.77, 95% CI 2-sided [-60.49 to -37.05], Standard Error of Mean 5.90 — Placebo is the reference
Statistical Analysis 3: Comparison: A20 Placebo Q2W vs A20 Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -52.68, 95% CI 2-sided [-64.06 to -41.30], Standard Error of Mean 5.73 — Placebo is the reference
Statistical Analysis 4: Comparison: A20 Placebo QM vs A20 Evolocumab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -39.97, 95% CI 2-sided [-50.46 to -29.48], Standard Error of Mean 5.29 — Placebo is the reference

19. Secondary Outcome: Percent Change From Baseline in Triglycerides at the Mean of Weeks 10 and 12
Time Frame: Baseline and Weeks 10 and 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | A5 Placebo Q2W | A5 Placebo QM | A5 Evolocumab Q2W | A5 Evolocumab QM | A20 Placebo Q2W | A20 Placebo QM | A20 Evolocumab Q2W | A20 Evolocumab QM
Number analyzed (Participants) | 49 | 50 | 50 | 50 | 52 | 51 | 51 | 51
percent change | 4.69 (6.04) | 4.54 (5.31) | -23.23 (6.15) | -17.41 (5.14) | -2.11 (4.45) | 8.06 (6.16) | -22.12 (4.44) | -12.66 (6.01)
Statistical Analysis 1: Comparison: A5 Placebo Q2W vs A5 Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -27.93, 95% CI 2-sided [-41.27 to -14.59], Standard Error of Mean 6.72 — Placebo is the reference
Statistical Analysis 2: Comparison: A5 Placebo QM vs A5 Evolocumab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -21.94, 95% CI 2-sided [-32.54 to -11.35], Standard Error of Mean 5.34 — Placebo is the reference
Statistical Analysis 3: Comparison: A20 Placebo Q2W vs A20 Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -20.01, 95% CI 2-sided [-29.59 to -10.43], Standard Error of Mean 4.83 — Placebo is the reference
Statistical Analysis 4: Comparison: A20 Placebo QM vs A20 Evolocumab QM; Test type: Superiority or Other; p = 0.010, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -20.72, 95% CI 2-sided [-34.18 to -7.26], Standard Error of Mean 6.78 — Placebo is the reference

20. Secondary Outcome: Percent Change From Baseline in Triglycerides at Week 12
Time Frame: Baseline and Week 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | A5 Placebo Q2W | A5 Placebo QM | A5 Evolocumab Q2W | A5 Evolocumab QM | A20 Placebo Q2W | A20 Placebo QM | A20 Evolocumab Q2W | A20 Evolocumab QM
Number analyzed (Participants) | 49 | 50 | 50 | 50 | 52 | 51 | 51 | 51
percent change | 7.84 (7.65) | 4.34 (5.61) | -19.73 (7.74) | -15.63 (5.43) | -3.88 (4.85) | 7.30 (6.42) | -21.05 (4.82) | -9.63 (6.26)
Statistical Analysis 1: Comparison: A5 Placebo Q2W vs A5 Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -27.57, 95% CI 2-sided [-46.33 to -8.81], Standard Error of Mean 9.45 — Placebo is the reference
Statistical Analysis 2: Comparison: A5 Placebo QM vs A5 Evolocumab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -19.97, 95% CI 2-sided [-31.68 to -8.25], Standard Error of Mean 5.90 — Placebo is the reference
Statistical Analysis 3: Comparison: A20 Placebo Q2W vs A20 Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -17.17, 95% CI 2-sided [-28.15 to -6.19], Standard Error of Mean 5.53 — Placebo is the reference
Statistical Analysis 4: Comparison: A20 Placebo QM vs A20 Evolocumab QM; Test type: Superiority or Other; p = 0.010, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -16.92, 95% CI 2-sided [-31.29 to -2.56], Standard Error of Mean 7.24 — Placebo is the reference

21. Secondary Outcome: Percent Change From Baseline in HDL-C at the Mean of Weeks 10 and 12
Time Frame: Baseline and Weeks 10 and 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | A5 Placebo Q2W | A5 Placebo QM | A5 Evolocumab Q2W | A5 Evolocumab QM | A20 Placebo Q2W | A20 Placebo QM | A20 Evolocumab Q2W | A20 Evolocumab QM
Number analyzed (Participants) | 49 | 50 | 50 | 50 | 52 | 51 | 51 | 51
percent change | -4.83 (2.25) | -1.57 (2.29) | 7.50 (2.30) | 13.05 (2.22) | -4.03 (2.34) | -3.06 (2.13) | 11.34 (2.33) | 6.09 (2.07)
Statistical Analysis 1: Comparison: A5 Placebo Q2W vs A5 Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = 12.33, 95% CI 2-sided [7.39 to 17.27], Standard Error of Mean 2.49 — Placebo is the reference
Statistical Analysis 2: Comparison: A5 Placebo QM vs A5 Evolocumab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = 14.61, 95% CI 2-sided [9.93 to 19.30], Standard Error of Mean 2.36 — Placebo is the reference
Statistical Analysis 3: Comparison: A20 Placebo Q2W vs A20 Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = 15.36, 95% CI 2-sided [10.12 to 20.60], Standard Error of Mean 2.64 — Placebo is the reference
Statistical Analysis 4: Comparison: A20 Placebo QM vs A20 Evolocumab QM; Test type: Superiority or Other; p = 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = 9.15, 95% CI 2-sided [4.67 to 13.62], Standard Error of Mean 2.26 — Placebo is the reference

22. Secondary Outcome: Percent Change From Baseline in HDL-C at Week 12
Time Frame: Baseline and Week 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | A5 Placebo Q2W | A5 Placebo QM | A5 Evolocumab Q2W | A5 Evolocumab QM | A20 Placebo Q2W | A20 Placebo QM | A20 Evolocumab Q2W | A20 Evolocumab QM
Number analyzed (Participants) | 49 | 50 | 50 | 50 | 52 | 51 | 51 | 51
percent change | -4.59 (2.58) | -0.40 (2.47) | 8.88 (2.62) | 14.80 (2.39) | -3.57 (2.59) | -2.36 (2.38) | 13.28 (2.58) | 7.84 (2.32)
Statistical Analysis 1: Comparison: A5 Placebo Q2W vs A5 Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = 13.46, 95% CI 2-sided [7.40 to 19.53], Standard Error of Mean 3.06 — Placebo is the reference
Statistical Analysis 2: Comparison: A5 Placebo QM vs A5 Evolocumab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = 15.20, 95% CI 2-sided [9.87 to 20.52], Standard Error of Mean 2.68 — Placebo is the reference
Statistical Analysis 3: Comparison: A20 Placebo Q2W vs A20 Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = 16.85, 95% CI 2-sided [10.74 to 22.95], Standard Error of Mean 3.08 — Placebo is the reference
Statistical Analysis 4: Comparison: A20 Placebo QM vs A20 Evolocumab QM; Test type: Superiority or Other; p = 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = 10.20, 95% CI 2-sided [4.85 to 15.55], Standard Error of Mean 2.70 — Placebo is the reference

23. Secondary Outcome: Percent Change From Baseline in VLDL-C at the Mean of Weeks 10 and 12
Time Frame: Baseline and Weeks 10 and 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | A5 Placebo Q2W | A5 Placebo QM | A5 Evolocumab Q2W | A5 Evolocumab QM | A20 Placebo Q2W | A20 Placebo QM | A20 Evolocumab Q2W | A20 Evolocumab QM
Number analyzed (Participants) | 49 | 50 | 50 | 50 | 52 | 51 | 51 | 51
percent change | 2.57 (5.52) | 3.10 (5.12) | -25.29 (5.65) | -19.55 (4.95) | -1.32 (4.32) | 9.96 (5.57) | -19.41 (4.31) | -17.20 (5.46)
Statistical Analysis 1: Comparison: A5 Placebo Q2W vs A5 Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -27.85, 95% CI 2-sided [-39.37 to -16.34], Standard Error of Mean 5.80 — Placebo is the reference
Statistical Analysis 2: Comparison: A5 Placebo QM vs A5 Evolocumab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -22.65, 95% CI 2-sided [-32.91 to -12.39], Standard Error of Mean 5.17 — Placebo is the reference
Statistical Analysis 3: Comparison: A20 Placebo Q2W vs A20 Evolocumab Q2W; Test type: Superiority or Other; p = 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -18.09, 95% CI 2-sided [-27.40 to -8.77], Standard Error of Mean 4.69 — Placebo is the reference
Statistical Analysis 4: Comparison: A20 Placebo QM vs A20 Evolocumab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -27.16, 95% CI 2-sided [-39.31 to -15.01], Standard Error of Mean 6.12 — Placebo is the reference

24. Secondary Outcome: Percent Change From Baseline in VLDL-C at Week 12
Time Frame: Baseline and Week 12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | A5 Placebo Q2W | A5 Placebo QM | A5 Evolocumab Q2W | A5 Evolocumab QM | A20 Placebo Q2W | A20 Placebo QM | A20 Evolocumab Q2W | A20 Evolocumab QM
Number analyzed (Participants) | 49 | 50 | 50 | 50 | 52 | 51 | 51 | 51
percent change | 4.09 (6.22) | 2.92 (5.45) | -24.33 (6.34) | -17.89 (5.27) | -3.03 (4.70) | 9.17 (5.63) | -18.08 (4.68) | -15.18 (5.52)
Statistical Analysis 1: Comparison: A5 Placebo Q2W vs A5 Evolocumab Q2W; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -28.42, 95% CI 2-sided [-42.48 to -14.36], Standard Error of Mean 7.08 — Placebo is the reference
Statistical Analysis 2: Comparison: A5 Placebo QM vs A5 Evolocumab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -20.81, 95% CI 2-sided [-32.29 to -9.33], Standard Error of Mean 5.78 — Placebo is the reference
Statistical Analysis 3: Comparison: A20 Placebo Q2W vs A20 Evolocumab Q2W; Test type: Superiority or Other; p = 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -15.05, 95% CI 2-sided [-25.72 to -4.39], Standard Error of Mean 5.37 — Placebo is the reference
Statistical Analysis 4: Comparison: A20 Placebo QM vs A20 Evolocumab QM; Test type: Superiority or Other; p < 0.001, Repeated measures linear effects model — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; [statistical method as in outcome 1, analysis 1]; LS Mean Treatment Difference = -24.35, 95% CI 2-sided [-36.70 to -11.99], Standard Error of Mean 6.22 — Placebo is the reference

ADVERSE EVENTS:
Time Frame: From the first dose of blinded investigational product until the end of the study (up to 14 weeks).
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | A5 Placebo Q2W | A5 Placebo QM | A5 Evolocumab Q2W | A5 Evolocumab QM | A20 Placebo Q2W | A20 Placebo QM | A20 Evolocumab Q2W | A20 Evolocumab QM
Serious Adverse Events (participants affected / at risk) | 1/49 | 2/50 | 0/50 | 1/50 | 1/52 | 1/51 | 0/51 | 0/51
Other Adverse Events (participants affected / at risk) | 11/49 | 11/50 | 13/50 | 9/50 | 6/52 | 14/51 | 7/51 | 12/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | A5 Placebo Q2W (N=49) | A5 Placebo QM (N=50) | A5 Evolocumab Q2W (N=50) | A5 Evolocumab QM (N=50) | A20 Placebo Q2W (N=52) | A20 Placebo QM (N=51) | A20 Evolocumab Q2W (N=51) | A20 Evolocumab QM (N=51)
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Brain stem infarction (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Epilepsy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | A5 Placebo Q2W (N=49) | A5 Placebo QM (N=50) | A5 Evolocumab Q2W (N=50) | A5 Evolocumab QM (N=50) | A20 Placebo Q2W (N=52) | A20 Placebo QM (N=51) | A20 Evolocumab Q2W (N=51) | A20 Evolocumab QM (N=51)
Gastroenteritis (Infections and infestations) | 1 | 0 | 1 | 2 | 1 | 0 | 0 | 3
Nasopharyngitis (Infections and infestations) | 10 | 10 | 12 | 7 | 5 | 11 | 7 | 8
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0 | 3 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.